CLINICAL TRIAL: NCT00852046
Title: Adjunct Dexmedetomidine Therapy Impact on Sedative and Analgesic
Brief Title: Adjunct Dexmedetomidine (Precedex®) Therapy Impact on Sedative and Analgesic Requirement
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI resigned.
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #2008.071
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-07

CONDITIONS: Sedation; Analgesia
Keywords: Mechanical ventilation
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. Low dose dexmedetomidine (Experimental): Dexmedetomidine 0.2 mcg/kg/hr added to fentanyl & propofol.
  Interventions: Drug: Dexmedetomidine
- 2. High dose dexmedetomidine (Experimental): Dexmedetomidine 0.6 mcg/kg/hr added to fentanyl & propofol.
  Interventions: Drug: Dexmedetomidine
- 3. Placebo (Placebo Comparator): Placebo added to fentanyl & propofol.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — IV solution, 0.2 mcg/kg/hr or 0.6 mcg/kg/hr for a max of 5 days
  Other Names: Precedex

SUMMARY:
Assess impact of increasing dose of dexmedetomidine on total daily dose of fentanyl and propofol while maintaining sedation in a mechanically ventilated patient in a general medical intensive care unit.

DETAILED DESCRIPTION:
Patients identified by selection criteria within 48 hours of intubation will be randomly assigned to one of three study arms: dexmedetomidine 0.2 mcg/kg/hr, dexmedetomidine 0.6 mcg/kg/hr, or placebo. If not already on, patients will be converted to propofol and fentanyl for sedation and analgesia, which will be titrated to a goal SAS score of 3-4.

Patients will be monitored, assessed, and evaluated by all regular policies and procedures of the institution. Extubation will be at the discretion of the physicians and medical team caring for the patient. If the patient is still intubated at five days study drug will then be stopped and further use of dexmedetomidine will be at the discretion of the physicians.

Primary objective will assess impact of increasing dose of dexmedetomidine on total daily dose of fentanyl and propofol while maintaining sedation in a mechanically ventilated patient in a general medical intensive care unit.

Secondary objectives include total ventilation time, ICU length of stay, hospital length of stay, patient outcomes/mortality, and total pharmacy expenditures.

ELIGIBILITY:
Inclusion Criteria:

* surgical, medical, or trauma patients requiring sedation for mechanical ventilation
* age 18-80
* Anticipated ventilation time of > 24 hrs
* Reasonable chance of recovery

Exclusion Criteria:

* Severe COPD
* Chronic immunosuppression (equivalent to prednisone 7.5 mg daily or higher)
* Heart block
* Bradycardia
* Significant head injury
* Goal SAS score of 1-2
* Severe hepatic impairment
* Hypertriglyceridemia
* Allergy to dexmedetomidine, fentanyl, propofol or eggs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Total daily dose of fentanyl and propofol | Daily

SECONDARY OUTCOMES:
Total ventilation time | Study ended
ICU length of stay | Study ended.
Hospital length of stay | Study ended
Patient outcomes/mortality | Study ended.
Total pharmacy expenditures | Study ended.

CONTACTS AND LOCATIONS:
Overall Officials: John A Kappes, Pharm.D., Principal Investigator — Avera McKennan Hospital